CLINICAL TRIAL: NCT05879510
Title: 68Ga-NY104 PET/CT for the Detection of Clear Cell Renal Cell Carcinoma in Presurgical Patients With Renal Masses
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCRPS
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: 68Ga-NY104; PET/CT; renal mass
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NY104 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-NY104 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NY104 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NY104 The recommended administered activity of 68Ga-NY104 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator.
  The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NY104 administration.
  Other Names: 68Ga-NYM005 PET/CT

SUMMARY:
This is a prospective, single-center, single-arm, diagnostic phase 2 study in patients who have renal masses scheduled for surgical resection. The goal is to determine the sensitivity and specificity of 68Ga-NY104 PET/CT in the detection of clear cell renal cell carcinoma using histopathological diagnosis as ground truth, in patients with operable renal masses.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, diagnostic phase 2 study in patients with renal masses scheduled for surgical resection. Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed. Additionally, prior to resection of the tumor, contrast-enhanced CT imaging of the abdomen, and if clinically warranted, or as part of the local standard of care, of the chest, will be performed. Both imaging modalities will be performed prior to resection of the kidney(s). PET/CT studies will be interpreted by two readers and diagnostic CT will be interpreted by one reader, all of whom will provide independent and blinded interpretations. Imaging interpretations and histopathologic evaluation data will be used to estimate the sensitivity, specificity, and predictive value (primary and secondary objectives) of each modality. The exploration into the detection of metastases by 68Ga-NY104 PET/CT in comparison to diagnostic CT will also be performed.

The pathologist will identify representative tumor tissue for the determination of histology, grading, and CAIX expression.

63 patients will be recruited in Peking Union Medical College Hospital. This study will be conducted according to local regulations and laws, the ethical principles that have their origin in the Declaration of Helsinki, and the principles of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Presence of a renal mass
3. Scheduled for surgical resection of renal mass (partial or total nephrectomy, open, laparoscopic, or robot-assisted technique)
4. Expected survival of at least 3 months
5. ECOG ≤ 2
6. Written informed consent provided for participation in the trial
7. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NY104 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NY104. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NY104 PET/CT is required.
2. Intercurrent medical condition that renders the patient ineligible for surgery.
3. Pregnancy or breastfeeding.
4. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Binary reading of renal lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  Define lesion as PET positive or PET negative lesion. The kidney lesion is designated as positive if the SUVmax of kidney lesions is higher than that of liver (reference).
Histological classification of operated renal lesions | From study completion to 1 month after completion
  The histological classification of operated renal lesions will be determined according to WHO classification of tumors, Feb 2004.

SECONDARY OUTCOMES:
SUVmax of renal lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  For kidney lesions, the tracer uptake is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimensional region of interest (ROI) over the lesion using a threshold of 40% SUVmax. The ROI should be drawn with caution not to include any adjacent normal kidney parenchyma.
SUVmax of liver uptake on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  The liver uptake (SUVmax (liver)) is used as the references to define PET positive lesions. It is measured by placing a 3-cm region of interest in right lobe at the level of porta hepatis. Focal lesion should be avoided if present.
Tumor grade of operated renal lesions | From study completion to 1 month after completion
  The tumor grade of operated renal lesions will be determined according to Fuhrmann grading system
Intensity of CAIX staining of operated renal lesions | From study completion to 1 month after completion
  The intensity of CAIX staining of operated renal lesions will be based on a 4-point scale from 0-3 according to the method of Bui et al, 2003
Extent of CAIX staining of operated renal lesions | From study completion to 1 month after completion
  The extent of CAIX staining of operated renal lesions will be determined by the percentage of the target tissue sample that have positive CAIX expression according to the method of Bui et al, 2003
Binary reading of renal lesions identified on diagnostic CT | From study completion to 1 month after completion
  A tumor will be described as clear cell renal carcinoma on a triphasic CT if one of the following two parameters is applicable:
  * Significant (>85 HU) enhancement in the cortico-medullary phase
  * Significant (>45 HU) enhancement in the parenchyma / excretory phase
Size of renal lesions identified on diagnostic CT | From study completion to 1 month after completion
  The longest diameter of the tumor will be measured on diagnostic CT
Number of metastatic lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NY104 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NY104 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Location of metastatic lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NY104 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NY104 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Szie of metastatic lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  For metastasis evaluation, any focal accumulation of 68Ga-NY104 outside the kidneys that cannot be explained by physiologic uptake is interpreted as focal lesion. The SUVmax and tumor-to-background should be evaluated. Surrounding tissue is the preferred background tissue. Should not available, the blood pool should be designated as background tissue. Any focal lesion identified on 68Ga-NY104 PET will be considered to be positive for metastasis if SUVmax (lesion) is no less than SUVmax (liver) or tumor-to-background ratio is higher than 1.
Number of metastatic lesions on diagnostic CT | From study completion to 1 month after completion
  The number of metastatic lesions on diagnostic CT will be determined by radiologist according to the typical location, enhancement pattern of the lesions.
Location of metastatic lesions on diagnostic CT | From study completion to 1 month after completion
  The number of metastatic lesions on diagnostic CT will be determined by radiologist according to the typical location, enhancement pattern of the lesions.
Size of metastatic lesions on diagnostic CT | From study completion to 1 month after completion
  The number of metastatic lesions on diagnostic CT will be determined by radiologist according to the typical location, enhancement pattern of the lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Within 2 years after the publication of the main results
Access Criteria: No limit.